CLINICAL TRIAL: NCT03905122
Title: Investigation of the Effects of Continuous Venous Dialysis and Hemodialysis on Fluid Dynamics by Bioreactance Method
Brief Title: Effects of Continuous Venous Dialysis and Hemodialysis on Fluid Dynamics by Bioreactance Method
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Prof Mehmet Turan Inal, Clinical Proffessor, Trakya University
Other Study IDs: TUTF-BAEK 2018/229
Record Dates: First submitted 2018-12-24; First posted 2019-04-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Renal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- continous veno-venous hemodialysis: to measure the fluid changes by using bioreactance method in continous veno-venous hemodialysis group
  Interventions: Device: bioreactans tool
- hemodialysis: to measure the fluid changes by using bioreactance method in hemodialysis group
  Interventions: Device: bioreactans tool

INTERVENTIONS:
Device: bioreactans tool — It is a completely non-invasive method by bioreactance method and it can be done to measure the intra-body fluid status with the help of the probes.

SUMMARY:
Dialysis methods applied at the bedside and dialysis methods applied in hemodialysis unit are widely applied in patients with renal insufficiency. Especially hemodynamically affected patients are less affected by hemodynamics as a result of using dialysis methods. It is a completely non-invasive method by bioreactance method and it can be done to measure the intra-body fluid status with the help of the glued probes. The aim of this study is to investigate the effects of continuous venous dialysis and hemodialysis on the fluid dynamics applied at the bedside with bioreactance method. In this way, the patient can develop more comfortable hemodynamic changes. Patients in the Surgery, Reanimation and Postoperative Intensive Care Unit with more than 24 hours of hospitalization and bedside dialysis or hemodialysis will be included in the study. Before the dialysis, body fluid measurements will be made with bioreactance, and after dialysis in patients receiving hemodialysis, and in dialysis patients 6, 12, 24 and 36 hours.

DETAILED DESCRIPTION:
Dialysis methods applied at the bedside and dialysis methods applied in hemodialysis unit are widely applied in patients with renal insufficiency. Especially hemodynamically affected patients are less affected by hemodynamics as a result of using dialysis methods. Dialysis in the hemodialysis unit is a method used in intensive care patients and is preferred especially in patients with stable hemodynamics. In dialysis methods, changes occur frequently in the body fluids of the patient. It is a completely non-invasive method by bioreactance method and it can be done to measure the intra-body fluid status with the help of the glued probes. The aim of this study is to investigate the effects of continuous venous dialysis and hemodialysis on the fluid dynamics applied at the bedside with bioreactance method. As a result of measurements with buioreactans method, fluid balance in patients will be understood more easily. In this way, the patient can develop more comfortable hemodynamic changes. Patients in the Surgery, Reanimation and Postoperative Intensive Care Unit with more than 24 hours of hospitalization and bedside dialysis or hemodialysis will be included in the study. Before the dialysis, body fluid measurements will be made with bioreactance, and after dialysis in patients receiving hemodialysis, and in dialysis patients 6, 12, 24 and 36 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients required dialysis therapy

Exclusion Criteria:

* under 18 years old
* confirmed or undiagnosed brain death

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of dialysis treatment
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
change in thoracic fluid content | before and after hemodialysis therapy, before bedside continous venovenous dialysis therapy and 6,12,24 and 36. hours
  change in thoracic fluid content
change in Cardiac Output | before and after hemodialysis therapy, before bedside continous venovenous dialysis therapy and 6,12,24 and 36. hours
  change in Cardiac Output
change in Cardiac Index | before and after hemodialysis therapy, before bedside continous venovenous dialysis therapy and 6,12,24 and 36. hours
  change in Cardiac Index
change in stroke volum | before and after hemodialysis therapy, before bedside continous venovenous dialysis therapy and 6,12,24 and 36. hours
  change in stroke volum

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Senol Uyar, Specialist, Principal Investigator — Trakya University, Edirne
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No